CLINICAL TRIAL: NCT06290219
Title: The Effect of Platelet-rich Plasma and Hyaluronic Acid Nasal Injection in the Treatment of Traumatic Olfactory Dysfunction
Brief Title: The Effect of Platelet-rich Plasma Nasal Injection in the Treatment of Traumatic Olfactory Dysfunction
Acronym: PRP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Rong-San Jiang, Professor, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF23509A
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Olfactory Nerve Injury With Anosmia (Diagnosis); Effect of Drug
MeSH Terms: conditions — Disease | interventions — Hyaluronic Acid; gluconic acid; Tablets; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet-rich plasma combined with hyaluronic acid nasal injection (Experimental): a nasal injection of platelet-rich plasma combined with hyaluronic acid at the first day of the treatment. At the same time, one tablet of zinc gluconate (10mg) three times a day for 12 weeks and traditional olfactory training with 4 separate bottles of phenyl ethyl alcohol, lemon, eucalyptus, and clove oil. Patients were told to sniff each odorant for 10 seconds, twice a day for 12 weeks.
  Interventions: Combination Product: platelet-rich plasma combined with hyaluronic acid; Drug: Zinc Gluconate 10 MG Oral Tablet; Device: 4 bottles of phenyl ethyl alcohol, lemon, eucalyptus, and clove oil
- Control (Active Comparator): one tablet of zinc gluconate (10mg) three times a day for 12 weeks and traditional olfactory training with 4 separate bottles of phenyl ethyl alcohol, lemon, eucalyptus, and clove. Patients were told to sniff each odorant for 10 seconds, twice a day for 12 weeks.
  Interventions: Drug: Zinc Gluconate 10 MG Oral Tablet; Device: 4 bottles of phenyl ethyl alcohol, lemon, eucalyptus, and clove oil

INTERVENTIONS:
Combination Product: platelet-rich plasma combined with hyaluronic acid — The project investigator injects plasma mixed with hyaluronic acid into the nasal septum and the medial side of the middle turbinate of the patient's nasal cavity under a nasal endoscope.
  Arms: platelet-rich plasma combined with hyaluronic acid nasal injection
Drug: Zinc Gluconate 10 MG Oral Tablet — one tablet three times a day for a period of 12 weeks
  Other Names: zinc tablet
Device: 4 bottles of phenyl ethyl alcohol, lemon, eucalyptus, and clove oil — Sniffing each odorant for 10 seconds, twice a day for 12 weeks

SUMMARY:
The purpose of this study is to explore the efficacy of injecting high-concentration platelet plasma combined with hyaluronic acid into the nasal olfactory mucosa in the treatment of traumatic anosmia.

DETAILED DESCRIPTION:
Causes of olfactory impairment include sinus diseases, post-viral olfactory dysfunction, neurological diseases, and post-traumatic lesions of the olfactory nerve. Since the outbreak of the COVID-19 in 2019, there has been a significant increase in the number of patients suffering from olfactory disorders, and the duration of loss of smell and taste varies. According to follow-up studies, nearly 46% of those patients still have symptoms of olfactory impairment one year after diagnosis, and nearly 7% have even completely lost their ability to smell. In recent years, injecting platelet-rich plasma into the nasal cavity has been a new method to improve the sense of smell. The effects of platelet-rich plasma can reduce chronic inflammation and cell-related damage and promote regeneration of olfactory tissue, while hyaluronic acid can promote the release of growth factors from platelets.

The purpose of this study is to explore the efficacy of injecting high-concentration platelet plasma combined with hyaluronic acid into the nasal olfactory mucosa in the treatment of traumatic anosmia. A total of 80 patients with olfactory dysfunction were collected from otolaryngology, head and neck outpatient clinics. Selection criteria are 18 years of age or older, and loss of olfactory function for more than 6 months after head trauma. Exclusion criteria are pregnant or lactating women, patients with compromised immune function, patients with acute or chronic sinus infection, patients with nasal polyps, patients with a history of sinonasal cancer, and patients with low platelets or hemophilia and other blood and blood cell-related diseases.

This study will establish experimental groups and control groups according to random distribution. Subjects in both groups received zinc tablets and olfactory training for 12 weeks. The experimental group additionally received an injection of platelet-rich plasma combined with hyaluronic acid. After treatment, patients return to the clinic to track the olfactory condition.

Before treatment, the subjects evaluated their olfactory function using a Visual Analogue Scale (VAS) and performed the phenyl ethyl alcohol odor detection threshold test and the traditional Chinese version of the University of Pennsylvania Olfactory Identification Test. In the experimental group, 10cc of blood will be drawn from the subjects in the experimental group, the drawn blood will be centrifuged, the centrifuge tube will be inverted 20 times to mix the plasma and hyaluronic acid, and finally 5cc of the plasma mixed with hyaluronic acid will be drawn out using an empty syringe. The project investigator injects plasma mixed with hyaluronic acid into the nasal septum and the medial side of the middle turbinate of the patient's nasal cavity under a nasal endoscope. The two groups will undergo the same olfactory tests three months later to compare the changes in olfactory function of the two groups of patients before and after treatment to explore the efficacy of injecting high-concentration platelet plasma combined with hyaluronic acid into the nasal olfactory mucosa to treat traumatic anosmia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, and loss of olfactory function for more than 6 months after head trauma

Exclusion Criteria:

* pregnant or lactating women, patients with compromised immune function, patients with acute or chronic sinus infection, patients with nasal polyps, patients with a history of sinonasal cancer, and patients with low platelets or hemophilia and other blood and blood cell-related diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
phenyl ethyl alcohol odor detection threshold test | up to 12 weeks
  The phenyl ethyl alcohol (PEA) odor detection threshold test uses a rose-like PEA odorant to assess a patient's odor detection threshold.
traditional Chinese version of University of Pennsylvania Smell Identification Test (TC-UPSIT) | up to 12 weeks
  TC-UPSIT is the traditional Chinese version of the University of Pennsylvania Smell Identification Test. It is a modified version of the North American version, with 8 unfamiliar odorants replaced by other odorants.29 The TC-UPSIT consists of 40 tests as it follows the North American version of the University of Pennsylvania Smell Identification Test. In each test, the brown strip at the bottom of the test page consists of microcapsules of an odorant, which is released by scratching the strip using a pencil tip. The patient sniffs the released odorant and selects a response from 4 odor descriptor options that are used to identify the odorant. The TC-UPSIT score is the number of correct responses among the 40 tests taken.

SECONDARY OUTCOMES:
Visual Analogue Scale | up to 12 weeks
  Before and after treatment, the subjects subjectively evaluated their olfactory function using a Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol
Time Frame: from January 1, 2027 to December 31, 2027
Access Criteria: Permission from the principal investigator
URL: https://www.vghtc.gov.tw

REFERENCES:
- [Background] Yan CH, Jang SS, Lin HC, Ma Y, Khanwalkar AR, Thai A, Patel ZM. Use of platelet-rich plasma for COVID-19-related olfactory loss: a randomized controlled trial. Int Forum Allergy Rhinol. 2023 Jun;13(6):989-997. doi: 10.1002/alr.23116. Epub 2022 Dec 21. PMID 36507615
- [Background] Steffens Y, Le Bon SD, Lechien J, Prunier L, Rodriguez A, Saussez S, Horoi M. Effectiveness and safety of PRP on persistent olfactory dysfunction related to COVID-19. Eur Arch Otorhinolaryngol. 2022 Dec;279(12):5951-5953. doi: 10.1007/s00405-022-07560-y. Epub 2022 Jul 29. PMID 35904632
- [Background] Lechien JR, Le Bon SD, Saussez S. Platelet-rich plasma injection in the olfactory clefts of COVID-19 patients with long-term olfactory dysfunction. Eur Arch Otorhinolaryngol. 2023 May;280(5):2351-2358. doi: 10.1007/s00405-022-07788-8. Epub 2022 Dec 15. PMID 36520209
- [Background] Goljanian Tabrizi A, Asadi M, Mohammadi M, Abedi Yekta A, Sohrabi M. Efficacy of Platelet-Rich Plasma as an Adjuvant Therapy to Endoscopic Sinus Surgery in Anosmia Patients with Sinonasal Polyposis: A Randomized Controlled Clinical Trial. Med J Islam Repub Iran. 2021 Nov 24;35:156. doi: 10.47176/mjiri.35.156. eCollection 2021. PMID 35341080
- [Background] AlRajhi B, Alrodiman OA, Alhuzali AF, Alrashed H, Alrodiman YA, Alim B. Platelet-rich plasma for the treatment of COVID-19 related olfactory dysfunction: a systematic review. Rhinology. 2023 Dec 1;61(6):498-507. doi: 10.4193/Rhin23.168. PMID 37772881
- See also: Institutional website — https://www.vghtc.gov.tw/
- Available data/document: Study Protocol — https://www.vghtc.gov.tw/ — Study Data/Document can be requested from the PI.